CLINICAL TRIAL: NCT04399538
Title: A PHASE 2A, 2-PART, RANDOMIZED, DOUBLE-BLIND, DOUBLE-DUMMY PLACEBO-CONTROLLED, PARALLEL-GROUP (SPONSOR OPEN) STUDY TO ASSESS PHARMACODYNAMICS AND SAFETY OF PF-06865571 (DGAT2I) COADMINISTERED WITH PF-05221304 (ACCI) IN ADULT PARTICIPANTS WITH PRESUMED NONALCOHOLIC STEATOHEPATITIS (NASH)
Brief Title: Study of Pharmacodynamics and Safety of DGAT2i and ACCi Coadministered in Participants With Sponsor-defined Presumed Non Alcoholic Steatohepatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: C3711005
Record Dates: First submitted 2020-05-20; First posted 2020-05-22 (Actual); Results first posted 2023-04-13 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-03

CONDITIONS: Nonalcoholic Steatohepatitis; Nonalcoholic Fatty Liver Disease
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — ervogastat

STUDY DESIGN:
Intervention Model Description: Dose-ranging of combination doses
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind, Double-dummy, Placebo controlled
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Placebo (Placebo Comparator): Participants will receive medication for 6 weeks
  Interventions: Drug: Placebo
- DGAT2i (25 mg BID) + ACCi (10 mg BID) (Experimental): Participants will receive medication for 6 weeks
  Interventions: Drug: PF-06865571; Drug: PF-05221304
- DGAT2i (100 mg BID) + ACCi (10 mg BID) (Experimental): Participants will receive medication for 6 weeks
  Interventions: Drug: PF-06865571; Drug: PF-05221304
- DGAT2i (300 mg QD) + ACCi (20 mg QD) (Experimental): Participants will receive medication for 6 weeks
  Interventions: Drug: PF-06865571; Drug: PF-05221304
- DGAT2i (300 mg BID) + ACCi (10 mg BID) (Experimental): Participants will receive medication for 6 weeks
  Interventions: Drug: PF-06865571; Drug: PF-05221304

INTERVENTIONS:
Drug: PF-06865571 — Tablet
  Other Names: DGAT2i
  Arms: DGAT2i (100 mg BID) + ACCi (10 mg BID); DGAT2i (25 mg BID) + ACCi (10 mg BID); DGAT2i (300 mg BID) + ACCi (10 mg BID); DGAT2i (300 mg QD) + ACCi (20 mg QD)
Drug: PF-05221304 — Tablet
  Other Names: ACCi
  Arms: DGAT2i (100 mg BID) + ACCi (10 mg BID); DGAT2i (25 mg BID) + ACCi (10 mg BID); DGAT2i (300 mg BID) + ACCi (10 mg BID); DGAT2i (300 mg QD) + ACCi (20 mg QD)
Drug: Placebo — Tablet
  Arms: Placebo

SUMMARY:
The study will evaluate the effect of coadministration of a range of doses of DGAT2i with 1 dose of ACCi, on hepatic steatosis and the ability of DGAT2i to mitigate ACCi-induced elevations in serum triglycerides. The study has a 2-part design with sequential conduct of Part 1 and Part 2 with each part conducted in distinct/separate cohorts of participants. The overall study design, objectives/endpoints, eligibility criteria for both parts is envisioned to be identical, however, data from Part 1 will be used to determine whether to conduct Part 2.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥25 and ≤ 40 kg/m2
* concomitant medical conditions associated with NAFLD

Exclusion Criteria:

* Evidence of other causes of liver disease such as Alcoholic steatohepatitis, (de)compensated cirrhosis, active viral hepatitis
* Any condition possibly affecting drug absorption
* Unstable liver function tests
* Recent cardiovascular event(s),
* Malignancies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2020-08-10 (Actual); Primary Completion 2022-03-31 (Actual); Study Completion 2022-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (19):
- United States (11):
  - Clinical Trials Research, Lincoln, California
  - Catalina Research Institute, LLC, Montclair, California
  - Excel Medical Clinical Trials, Boca Raton, Florida
  - Optimus U Corporation, Miami, Florida
  - Floridian Clinical Research, LLC, Miami Lakes, Florida
  - East-West Medical Research Institute, Honolulu, Hawaii
  - L-MARC Research Center, Louisville, Kentucky
  - The Christ Hospital, Cincinnati, Ohio
  - Sterling Research Group, Ltd., Cincinnati, Ohio
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - National Clinical Research, Inc., Richmond, Virginia
- Canada (8):
  - Nova Scotia Health Authority QE II Health Sciences Centre, Halifax, Nova Scotia
  - Nova Scotia Health Authority - Queen Elizabeth II Health Sciences Centre, Halifax, Nova Scotia
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Milestone Research Inc., London, Ontario
  - Resonance Magnetique du Saguenay-Lac-Saint-Jean, Chicoutimi, Quebec
  - Ecogene-21, Chicoutimi, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
  - Centre de Recherche Saint-Louis, Québec

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3711005

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In Part 1, 76 participants were enrolled and 75 were randomized (including 1 participant who was randomized 2 times at the same site), and 74 unique participants received at least 1 dose of study intervention. A decision was made that Part 2 would not proceed based on Part 1 interim analysis, therefore enrollment for Part 2 was not conducted.
Groups:
- Placebo: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. Each dose contained 2 large tablets (placebo tablets matching the diacylglycerol acyltransferase 2 inhibitor [DGAT2i] PF-06865571) plus 1 small tablet (placebo tablet matching the acetyl-CoA carboxylase inhibitor [ACCi] PF-05221304). Two follow-up visits were scheduled after end of treatment.
- PF-06865571 25 mg Twice Daily (BID) + PF-05221304 10 mg BID: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. Each dose contained 2 large tablets (1 DGAT2i-matching placebo tablet, 1 DGAT2i 25 mg tablet) plus 1 small tablet (ACCi 10 mg tablet). Two follow-up visits were scheduled after end of treatment.
- PF-06865571 100 mg BID + PF-05221304 10 mg BID: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. Each dose contained 2 large tablets (2 DGAT2i 50 mg tablets) plus 1 small tablet (ACCi 10 mg tablet). Two follow-up visits were scheduled after end of treatment. Two follow-up visits were scheduled after end of treatment.
- PF-06865571 300 mg Once Daily (QD) + PF-05221304 20 mg QD: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. The morning dose contained 2 large tablets (2 DGAT2i 150 mg tablets) plus 1 small tablet (ACCi 20 mg tablet). The evening dose contained 2 large tablets (2 DGAT2i-matching placebo tablets) plus 1 small tablet (ACCi-matching placebo tablet). Two follow-up visits were scheduled after end of treatment.
- PF-06865571 300 mg BID + PF-05221304 10 mg BID: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. Each dose contained 2 large tablets (2 DGAT2i 150 mg tablets) plus 1 small tablet (ACCi 10 mg tablet). Two follow-up visits were scheduled after end of treatment.
Period: Double-Blind Treatment
Arm/Group | Placebo | PF-06865571 25 mg Twice Daily (BID) + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg Once Daily (QD) + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Started | 15 | 15 | 13 | 18 | 14
Completed | 15 | 15 | 13 | 17 | 12
Not Completed | 0 | 0 | 0 | 1 | 2
Not completed — Work schedule conflicts | 0 | 0 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Period: Follow-Up
Arm/Group | Placebo | PF-06865571 25 mg Twice Daily (BID) + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg Once Daily (QD) + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Started | 15 | 15 | 13 | 17 | 13
Completed | 15 | 15 | 13 | 15 | 12
Not Completed | 0 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Baseline population included all participants who were randomized and received at least 1 dose of study intervention.
Groups:
- PF-06865571 25 mg BID + PF-05221304 10 mg BID: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. Each dose contained 2 large tablets (1 DGAT2i-matching placebo tablet, 1 DGAT2i 25 mg tablet) plus 1 small tablet (ACCi 10 mg tablet). Two follow-up visits were scheduled after end of treatment.
- PF-06865571 100 mg BID + PF-05221304 10 mg BID: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. Each dose contained 2 large tablets (2 DGAT2i 50 mg tablets) plus 1 small tablet (ACCi 10 mg tablet). Two follow-up visits were scheduled after end of treatment.
- PF-06865571 300 mg QD + PF-05221304 20 mg QD: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. The morning dose contained 2 large tablets (2 DGAT2i 150 mg tablets) plus 1 small tablet (ACCi 20 mg tablet). The evening dose contained 2 large tablets (2 DGAT2i-matching placebo tablets) plus 1 small tablet (ACCi-matching placebo tablet). Two follow-up visits were scheduled after end of treatment.
- Total: Total of all reporting groups
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID | Total
Number analyzed (Participants) | 15 | 15 | 13 | 18 | 13 | 74
Age, Continuous [Median (Full Range); unit: Years] | 57.00 [33 to 72] | 54.00 [35 to 69] | 56.00 [43 to 66] | 50.00 [25 to 72] | 56.00 [32 to 69] | 54.50 [25 to 72]
Age, Customized [Count of Participants; unit: Participants]
  18-44 years | 3 | 2 | 1 | 3 | 4 | 13
  45-64 years | 10 | 11 | 9 | 12 | 7 | 49
  >=65 years | 2 | 2 | 3 | 3 | 2 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 8 | 7 | 7 | 4 | 34
  Male | 7 | 7 | 6 | 11 | 9 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 9 | 8 | 9 | 4 | 38
  Not Hispanic or Latino | 7 | 6 | 5 | 9 | 9 | 36
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 3 | 4 | 1 | 4 | 1 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 0 | 1 | 2
  White | 12 | 11 | 11 | 14 | 11 | 59
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline (CFB) in Percent (%) Liver Fat as Assessed Via Magnetic Resonance Imaging Using Proton Density Fat Fraction Acquisition (MRI-PDFF) at Week 6
Description: MRI-PDFF technique is an established method that enables quantification of fat content in the liver. It measures the fraction of mobile protons in the liver attributable to fat content and provides whole liver coverage so that fat content can be assessed across 8 Couinaud liver segments. Whole liver PDFF = the sum of PDFFs for (Segment I + Segment II + Segment III + Segment IVa + Segment IVb + Segment V + Segment VI + Segment VII + Segment VIII) divided by (number of segments assessed and no missing/mapping at Baseline, and on Week 6). If some segments did not have results reported at Baseline and/or Week 6, liver PDFF was to be calculated using data in segments that had data available at both Baseline visit and Week 6 visit. For this outcome measure (OM), baseline is defined as the assessment undertaken between Visit 3/Week -2 and Visit 4/Day 1.
Time Frame: Baseline, Week 6
Population: The analysis population included all participants randomized who received at least 1 dose of study intervention (Placebo/DGAT2i + ACCi), and had at least 1 observation in the model used for this OM.
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Number analyzed (Participants) | 15 | 14 | 12 | 13 | 9
Percent change | -3.58 [-14.71 to 8.99] | -54.07 [-59.54 to -47.85] | -58.14 [-63.51 to -51.98] | -60.28 [-65.27 to -54.57] | -47.75 [-55.71 to -38.35]
Statistical Analysis 1: Comparison: Placebo vs PF-06865571 25 mg BID + PF-05221304 10 mg BID; Natural log-transformed individual relative change (RC) from baseline to Week 6 was analyzed using the ANCOVA model with treatment as a fixed effect, natural log-transformed baseline % liver fat by MRI-PDFF as covariate. Values were back-transformed from the log scale; Test type: Superiority; p < 0.0001, ANCOVA; Difference in least square (LS) mean = -52.36, 80% CI [-60.07 to -43.17]
Statistical Analysis 2: Comparison: Placebo vs PF-06865571 100 mg BID + PF-05221304 10 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS mean = -56.58, 80% CI [-63.88 to -47.80]
Statistical Analysis 3: Comparison: Placebo vs PF-06865571 300 mg QD + PF-05221304 20 mg QD; Natural log-transformed individual relative change (RC) from baseline to Week 6 was analyzed using the ANCOVA model with treatment as a fixed effect, natural log-transformed baseline % liver fat by MRI-PDFF as covariate. Values were back-transformed from the log scale. Relative change was converted to percent change as follows: Percent change = 100*(RC-1). 80% CI was calculated based on difference in LS mean between groups; Test type: Superiority; p < 0.0001, ANCOVA; Difference in LS mean = -58.80, 80% CI [-65.66 to -50.57]
Statistical Analysis 4: Comparison: Placebo vs PF-06865571 300 mg BID + PF-05221304 10 mg BID; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.0003, ANCOVA; Difference in LS mean = -45.80, 80% CI [-55.86 to -33.46]

2. Secondary Outcome: Percent CFB in Fasting Serum Triglycerides at Week 6
Description: Blood samples were collected before morning dose for the measurement of fasting serum triglycerides. Natural log transformed relative changes from baseline in fasting serum triglycerides were analyzed using mixed model repeated measures (MMRM) analysis with treatment, week and treatment by-week interaction as fixed effects, participant as random effect and log transformed baseline as a covariate using unstructured covariance structure. Values were back-transformed from the log scale. Relative change was converted to percent change as follows: Percent change = 100*(RC-1). For this OM, baseline is defined as the result closest prior to dosing on Day 1 (either predose on Day 1/Visit 4 or Week -2/Visit 3).
Time Frame: Baseline, Week 6
Population: as for outcome 1
Measure: Least Squares Mean (80% Confidence Interval); unit: Percent change
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Number analyzed (Participants) | 15 | 15 | 13 | 17 | 10
Percent change | 3.72 [-6.90 to 15.55] | 27.89 [14.75 to 42.53] | 18.00 [5.10 to 32.49] | 24.88 [12.85 to 38.20] | 14.69 [0.59 to 30.78]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=all AEs included in the AE Case Report Form (CRF) page during the study. A serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life threatening; required inpatient hospitalization or prolongation of existing hospitalization; resulted in persistent or significant disability/incapacity; or resulted in congenital anomaly/birth defect. Severe TEAEs were defined as AEs that prevent normal everyday activities. Treatment-related TEAEs were determined by the investigator.
Time Frame: Baseline up to at least 28 days after the last administration of the study intervention or until study completion or withdrawal, whichever was longer (maximum of approximately 24 weeks).
Population: The analysis population included all participants who were randomized to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Number analyzed (Participants) | 15 | 15 | 13 | 18 | 14
Participants
  All-causality TEAE | 2 | 4 | 5 | 6 | 7
  Treatment-related TEAE | 0 | 0 | 3 | 2 | 3
  SAE | 0 | 0 | 0 | 0 | 0
  All-causality severe TEAE | 0 | 0 | 0 | 1 | 0
  Treatment-related severe TEAE | 0 | 0 | 0 | 1 | 0
  All-causality TEAE leading to discontinuation from study | 0 | 0 | 0 | 0 | 1
  Treatment-related TEAE leading to discontinuation from study | 0 | 0 | 0 | 0 | 1

4. Secondary Outcome: Number of Participants With TEAEs of Special Interest by Preferred Term (PT)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship with study treatment. TEAEs=all AEs included in the AE CRF page during the study. A 3-tier approach was used to summarize and classify TEAEs into 1 of 3 tiers by the investigator based on their incidence rate and clinical importance to the trial. Tier-1 events = pre-specified events of clinical importance that are maintained in a program level list. Tier-2 events = events that are not tier-1 but are "common". A Medical Dictionary for Regulatory Activities Terminology (MedDRA) PT is defined as a tier-2 event if there are at least 4 participants with at least one occurrence in any treatment group, to distinguish Tier-2 events from Tier-3 events. Tier-3 events = events that do not meet criteria for either tier-1 or tier-2 event. TEAE(s) of special interest reported in at least 1 participant are presented in this OM.
Time Frame: as for outcome 3
Population: The analysis population included all participants who were randomized to study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Number analyzed (Participants) | 15 | 15 | 13 | 18 | 14
Participants
  Tier-1: Thrombocytopenia | 0 | 0 | 0 | 1 | 0
  Tier-1: Hypertriglyceridaemia | 0 | 0 | 0 | 1 | 0

5. Secondary Outcome: Number of Participants With Laboratory Test Abnormalities Without Regard to Baseline Abnormality
Description: Participants with laboratory test abnormalities (hematology, chemistry and urinalysis) meeting pre-specified criteria are reported without regard to baseline abnormality. LLN is lower limit of normal. ULN is upper limit of normal. Baseline was defined as the result closest prior to Day 1 dosing.
Time Frame: From baseline to end of follow-up or until study discontinuation/withdrawal, whichever was longer (maximum of approximately 19 weeks)
Population: The analysis population included all participants who were randomized and received at least 1 dose of study intervention. Number of participants analyzed = number of participants evaluable for this OM. Number analyzed = number of participants evaluable for each category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Number analyzed (Participants) | 15 | 15 | 13 | 18 | 13
Participants
  Hematology: Erythrocytes <0.8 x LLN | 0 | 0 | 0 | 1 | 0
  Hematology: Erythrocytes Mean Corpuscular Volume <0.9 x LLN | 1 | 0 | 0 | 0 | 0
  Hematology: Erythrocytes Mean Corpuscular Hemoglobin <0.9 x LLN | 0 | 2 | 0 | 0 | 0
  Hematology: Lymphocytes >1.2 x ULN | 0 | 0 | 0 | 0 | 1
  Hematology: Basophils >1.2 x ULN | 0 | 0 | 0 | 0 | 1
  Hematology: Eosinophils >1.2 x ULN | 0 | 1 | 0 | 1 | 1
  Clinical chemistry: Bicarbonate >1.1 X ULN | 0 | 0 | 1 | 0 | 0
  Clinical chemistry: Creatine kinase >2.0 X ULN | 0 | 0 | 1 | 0 | 1
  Urinalysis: Urine glucose >=1 | 2 | 1 | 1 | 3 | 2
  Urinalysis: Ketones >=1 | 0 | 0 | 2 | 2 | 2
  Urinalysis: Urine protein >=1 | 0 | 0 | 0 | 0 | 1
  Urinalysis: Urine hemoglobin | 0 | 0 | 0 | 1 | 0
  Urinalysis: Urobilinogen >=1 | 0 | 0 | 0 | 1 | 0
  Urinalysis: Nitrite >=1 | 2 | 1 | 0 | 1 | 1
  Urinalysis: Leukocyte Esterase >=1 | 5 | 3 | 3 | 4 | 3
  Urinalysis: Urine leukocytes (/high power field [HPF]) >=20: number analyzed (Participants) | 8 | 8 | 10 | 14 | 6
  Urinalysis: Urine leukocytes (/high power field [HPF]) >=20 | 2 | 0 | 0 | 0 | 1
  Urinalysis: Hyaline Casts (/low power field [LPF]) >1: number analyzed (Participants) | 2 | 1 | 0 | 2 | 0
  Urinalysis: Hyaline Casts (/low power field [LPF]) >1 | 2 | 0 | 0 | 0 | 0

6. Secondary Outcome: Number of Participants With Abnormalities in Laboratory Parameters of Special Interest Meeting Pre-Defined Criteria
Description: Laboratory parameters of special interest included fasting serum triglycerides, platelet count, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, total bilirubin, direct bilirubin, and fasting plasma glucose. Pre-specified criteria for laboratory parameters of special interest included flag level threshold (reflecting either the threshold for study entry or clinical significance) and alert level threshold (requiring rapid notification to site and study team when values exceeding the threshold were noted during the study). All flag level changes and alert level changes were cumulative from baseline (defined as result closest prior to dosing at Day 1). LLN is lower limit of normal. ULN is upper limit of normal.
Time Frame: as for outcome 5
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Number analyzed (Participants) | 15 | 15 | 13 | 18 | 13
Participants
  Platelet count <100x10^3/mm^3 (flag level) | 0 | 0 | 0 | 0 | 0
  Platelet count <75x10^3/mm^3 (alert level) | 0 | 0 | 0 | 0 | 0
  Bilirubin >1.5xULN (flag level) | 0 | 0 | 0 | 0 | 0
  Bilirubin >3xULN (alert level) | 0 | 0 | 0 | 0 | 0
  Direct bilirubin >ULN (flag level) | 0 | 0 | 0 | 0 | 0
  Aspartate aminotransferase >= 2xULN (flag level) | 0 | 4 | 4 | 5 | 3
  Aspartate aminotransferase >3xULN (flag level) | 0 | 1 | 0 | 1 | 0
  Aspartate aminotransferase >5xULN (flag level) | 0 | 1 | 0 | 0 | 0
  Aspartate aminotransferase >8xULN (alert level) | 0 | 0 | 0 | 0 | 0
  Alanine aminotransferase >=2xULN (flag level) | 4 | 6 | 7 | 6 | 4
  Alanine aminotransferase >3xULN (flag level) | 0 | 3 | 1 | 3 | 2
  Alanine aminotransferase >5xULN (flag level) | 0 | 1 | 0 | 0 | 0
  Alanine aminotransferase >8xULN (alert level) | 0 | 1 | 0 | 0 | 0
  Gamma glutamyl transferase >ULN (flag level) | 6 | 7 | 9 | 10 | 4
  Alkaline phosphatase >=2xULN (flag level) | 0 | 0 | 1 | 0 | 0
  Alkaline phosphatase >3xULN (flag level) | 0 | 0 | 0 | 0 | 0
  Alkaline phosphatase >5xULN (flag level) | 0 | 0 | 0 | 0 | 0
  Fasting plasma glucose <70 mg/dL (flag level): number analyzed (Participants) | 15 | 15 | 13 | 18 | 12
  Fasting plasma glucose <70 mg/dL (flag level) | 0 | 0 | 0 | 0 | 0
  Fasting plasma glucose >=140 mg/dL (flag level): number analyzed (Participants) | 15 | 15 | 13 | 18 | 12
  Fasting plasma glucose >=140 mg/dL (flag level) | 4 | 4 | 4 | 9 | 2
  Fasting plasma glucose <=49 mg/dL (alert level): number analyzed (Participants) | 15 | 15 | 13 | 18 | 12
  Fasting plasma glucose <=49 mg/dL (alert level) | 0 | 0 | 0 | 0 | 0
  Fasting plasma glucose >270 mg/dL (alert level): number analyzed (Participants) | 15 | 15 | 13 | 18 | 12
  Fasting plasma glucose >270 mg/dL (alert level) | 0 | 0 | 0 | 1 | 0
  Fasting serum triglycerides >=400 mg/dL (flag level): number analyzed (Participants) | 15 | 15 | 13 | 18 | 12
  Fasting serum triglycerides >=400 mg/dL (flag level) | 1 | 0 | 3 | 4 | 1
  Fasting serum triglycerides >=600 mg/dL (alert level): number analyzed (Participants) | 15 | 15 | 13 | 18 | 12
  Fasting serum triglycerides >=600 mg/dL (alert level) | 1 | 0 | 0 | 1 | 0
  Fasting serum triglycerides >=800 mg/dL (alert level): number analyzed (Participants) | 15 | 15 | 13 | 18 | 12
  Fasting serum triglycerides >=800 mg/dL (alert level) | 0 | 0 | 0 | 0 | 0

7. Secondary Outcome: Number of Participants With Post-Baseline Vital Signs Data Meeting Pre-Defined Criteria
Description: Pre-defined categorical criteria for vital signs data of special clinical concern included: seated systolic blood pressure (BP) absolute value <90 mmHg or change from baseline >=30 mmHg, seated diastolic BP absolute value <50 mmHg or change from baseline >=20 mmHg, seated pulse rate absolute value <40 beats per minute (bpm) or >120 bpm. Baseline was defined as the result closest prior to Day 1 dosing.
Time Frame: Baseline, Week 6, the first follow-up visit (Week 8), and the date of discontinuation/withdrawal from study (maximum of approximately 12 weeks after Day 1) if applicable
Population: The analysis population included all participants randomized who received at least 1 dose of study intervention and were evaluable for vital signs.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Number analyzed (Participants) | 15 | 15 | 13 | 18 | 13
Participants | 0 | 0 | 0 | 1 | 0

8. Secondary Outcome: Number of Participants With Post-Baseline Electrocardiogram (ECG) Data Meeting Pre-Defined Criteria
Description: Pre-defined categorical criteria for ECG data of special clinical concern included: (1) QTc interval absolute value >450 and <=480 msec (mild prolongation), >480 and <=500 msec (moderate prolongation), >500 msec (severe prolongation); (2) QTc interval increase from baseline >=30 and <=60 msec (moderate prolongation), or >60 msec (severe prolongation); (3) uncorrected QT interval >500 msec. ECG abnormalities meeting prespecified criteria and reported in at least 1 participant are presented in this OM. Baseline was defined as the result closest prior to Day 1 dosing.
Time Frame: as for outcome 7
Population: The analysis population included all participants randomized who received at least 1 dose of study intervention and were evaluable for ECG.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
Number analyzed (Participants) | 15 | 15 | 13 | 18 | 13
Participants
  450 msec <= QTc interval <480 msec | 1 | 0 | 0 | 0 | 1
  30 msec <= change from baseline in QTc interval <60 msec | 1 | 1 | 1 | 1 | 0
  change from baseline in QTc interval >=60 msec | 0 | 0 | 0 | 0 | 1

ADVERSE EVENTS:
Time Frame: Baseline up to at least 28 days after the last administration of the study intervention or until study completion or withdrawal, whichever was longer (maximum of approximately 24 weeks).
Description: The same event may appear as both an AE and an SAE. An event may be categorized as serious in one participant and as non-serious in another participant, or one participant may have experienced both a serious and non-serious event during the study. Total number at risk below refers to the number of participants evaluable for SAEs or AEs.
Groups:
- PF-06865571 25 mg BID + PF-05221304 10 mg BID: Participants had 2 oral doses per day (1 dose with the morning meal and 1 dose with the evening meal) for up to 6 weeks. Each dose contained 2 large tablets (1 DGAT2i-matching placebo tablet, 1 DGAT2i 25 mg tablet) plus 1 small tablet (ACCi 10 mg tablet). Two follow-up visits were scheduled after end of treatment. Two follow-up visits were scheduled after end of treatment.
Arm/Group | Placebo | PF-06865571 25 mg BID + PF-05221304 10 mg BID | PF-06865571 100 mg BID + PF-05221304 10 mg BID | PF-06865571 300 mg QD + PF-05221304 20 mg QD | PF-06865571 300 mg BID + PF-05221304 10 mg BID
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 0/18 | 0/14
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/13 | 0/18 | 0/14
Other Adverse Events (participants affected / at risk) | 2/15 | 4/15 | 5/13 | 6/18 | 7/14
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | PF-06865571 25 mg BID + PF-05221304 10 mg BID (N=15) | PF-06865571 100 mg BID + PF-05221304 10 mg BID (N=13) | PF-06865571 300 mg QD + PF-05221304 20 mg QD (N=18) | PF-06865571 300 mg BID + PF-05221304 10 mg BID (N=14)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0 | 2 | 1
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 0 | 1
Vaccination site pain (General disorders) | 0 | 0 | 1 | 0 | 0
Gastrointestinal viral infection (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Chest injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 1 | 0
Cytokeratin 18 increased (Investigations) | 0 | 0 | 0 | 1 | 0
SARS-CoV-2 antibody test positive (Investigations) | 0 | 0 | 0 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 0 | 0 | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Crystalluria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2020-03-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT04399538/Prot_000.pdf
  • Statistical Analysis Plan (2021-06-16): https://cdn.clinicaltrials.gov/large-docs/38/NCT04399538/SAP_001.pdf